CLINICAL TRIAL: NCT06721702
Title: The Effect of Motivational Interviewing on Internet Addiction and Digital Game Addiction in Adolescents
Brief Title: Motivational Interviewing and Addiction
Acronym: MI-IA-DGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ayaz Alkaya, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09.05.2023-757
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-12

CONDITIONS: Internet Addiction; Game Addiction, Video
Keywords: motivational interviewing; Adolescent; digital game addiction; problematic internet use
MeSH Terms: conditions — Internet Addiction Disorder; Technology Addiction | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: Motivational Interviewing (Experimental): The motivational interview, consisting of six sessions, including the preparation session, was applied to the intervention group.Each session lasted an average of 40 minutes. Motivational interviewing sessions were conducted with nine different groups consisting of five people in the intervention group.
  Interventions: Behavioral: Motivational interviewing
- Control Group (No Intervention): Control group did not receive any intervention other than the daily routine practices.

INTERVENTIONS:
Behavioral: Motivational interviewing — Motivational interviews were administered as the intervention of the research. Motivational interviewing consists of two stages. In the first stage, the four principles of motivational interviewing (developing contradiction, showing empathy, supporting self-efficacy, and resolving resistance) are aimed at providing motivation in individuals. The second stage is strengthening the commitment to change.
  Arms: Intervention group: Motivational Interviewing

SUMMARY:
The increasing use of the internet makes understanding games among adolescents different by moving it to the virtual environment and increases the digital game addiction risk. Especially among adolescents, digital games have become a popular activity and often a means of socialization. With the widespread use of smartphones, digital gaming has transformed from computer and console-based to a multi-platform activit. In addition, long-term digital games cause symptoms such as anxiety and depression through increased interpersonal loneliness and decreased relationships. This situation has caused recent research to focus on the effects of digital gaming activities on individuals.

DETAILED DESCRIPTION:
Internet addiction and digital game addiction, which are the negative side of rapidly developing digital technologies and increasing internet accessibility, are of global concern. Therefore, implementing interventions for internet and digital game addiction can be an effective approach to prevent physical, mental, environmental, and social problems caused by addiction. In this context, it is predicted that motivational interviewing may be an appropriate approach in combating internet and digital game addiction. Motivational interviewing is a client-centered psychotherapeutic approach that helps the person with ambivalence make positive decisions, achieve specific and better goals, and increase internal motivation for change. It is thought that motivational interviewing could contribute to reducing addictive behaviors by evaluating the effect of motivational interviewing on both internet addiction and digital game addiction at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Being a ninth-grade student
* Being in the intention or pre-intention stage according the change assessment form
* Being addicted to digital games
* Having family approval
* Volunteering to participate in the research

Exclusion Criteria:

• Having any physical and mental illness

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — To ensure homogeneity between the groups, gender was taken into consideration. Adolescents were divided into two strata according to gender (girls, boys), and allocated to experimental and control group at ratio 1:1.
Enrollment: 88 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Internet Addiction | 6 months up to July 2024
  Internet Addiction Test Short Form (YIBT-SF) was developed by Young (1998). It was converted into a short form by Pawlikowski et al (2013). It is a 5-point Likert-type scale consisting of 12 items and a single factor adapted into Turkish by Kutlu et al. in 2016. The scores obtained from the scale vary between 12 and 60. High scores obtained from the scale indicate a high level of dependency.
  The Cronbach's alpha coefficient obtained in the reliability study was found to be 0.86 in adolescents.
Digital Game Addiction | 6 months up to July 2024
  The Digital Game Addiction Scale (DGAS) was developed by Lemmens et al. (2009) to determine the problematic digital game playing behaviors of adolescents aged 12 - 18 years. The scale is a seven-item short form of the DGAS - 21, consisting of 21 items and seven sub-dimensions. The validity and reliability study of the Turkish version of the scale was conducted by Irmak and Erdoğan (2015). The validity and reliability values of the original DGAS were 0.92 for Cronbach 's alpha. The assessment is made using monoethic and polyethic diagnoses. According to the monothetic diagnosis, a person is defined as "game addicted" if they score three (sometimes) or more on all seven items; according to the polyethic diagnosis, a person is defined as "game addicted" if they score three (sometimes) or more on at least four of the seven items.

CONTACTS AND LOCATIONS:
Locations (1):
- Şehit Muhammet Onur Demir Anadolu High School, Halis Gülle Anadolu High School, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang YS, Liu TH, Qin D, Wang ZP, He XY, Chen YN. Effects of non-pharmacological interventions on youth with internet addiction: a systematic review and meta-analysis of randomized controlled trials. Front Psychiatry. 2024 Jan 11;14:1327200. doi: 10.3389/fpsyt.2023.1327200. eCollection 2023. PMID 38274427